CLINICAL TRIAL: NCT04495712
Title: Antiarrhythmic Effects of Spironolactone in Patients With ICDs
Acronym: SPIRIT
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ICDAD-1; VA 02-2704 (Other Grant/Funding Number: Department of Defene and VA)
Record Dates: First submitted 2020-07-28; First posted 2020-08-03 (Actual); Results first posted 2020-09-04 (Actual); Last update posted 2020-10-09 (Actual); Status verified 2020-10

CONDITIONS: Ventricular Arrhythmias
Keywords: Anti-Arrhythmia Agents; Ventricular Fibrillation; Ventricular Tachycardia; Defibrillators, Implantable
MeSH Terms: conditions — Ventricular Fibrillation; Tachycardia, Ventricular | interventions — Spironolactone

STUDY DESIGN:
Intervention Model Description: This was a prospective, double-blind, randomized trial that assigned patients to receive either spironolactone 25 mg/day or a placebo.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: All participants, providers, investigators, and outcome assessors were blinded to treatment assignment. The pharmacy maintained a key to randomization that was not broken until the study was completed and all outcomes had been assessed.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Spironolactone (Active Comparator): Patients randomized to active therapy with spironolactone
  Interventions: Drug: spironolactone
- placebo (Placebo Comparator): patients randomized to placebo
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: spironolactone — aldosterone blocker
  Other Names: Aldactone
  Arms: Spironolactone
Drug: placebo — identical in appearance to spironolactone study drug
  Arms: placebo

SUMMARY:
This study will test whether spironolactone, an approved drug for among other things hypertension, will reduce the risk of severe arrhythmias in patients with implanted defibrillators. Half the patients in the study will get spironolactone and half will get a placebo. Neither the patients or their providers will know if they are getting spironolactone or placebo.

DETAILED DESCRIPTION:
Objectives: This study is designed to determine whether spironolactone at a dose of 25 mg per day in patients with implanted cardioverter defibrillators (ICD) will 1) Reduce the incidence of ventricular tachycardia (VT) and ventricular fibrillation (VF), 2) Improve health related quality of life, 3) Reduce the need for hospitalization, and 4) Change ventricular refractoriness.

Plan: The study was a randomized double blind placebo controlled multi-center trial. Patients were randomized to either 25 mg per day of spironolactone or placebo and followed for 2 years each. The primary endpoint is time to the first episode of VT/VF. Secondary endpoints will include changes in health related quality of life, frequency of hospitalization, and in a subset of patients the effect of spironolactone on the ventricular effective refractory period measured through the ICD 3 months after starting the study medication. All data analyses will be conducted on intent to treat basis.

Methods: Patients were recruited at the Portland VA ICD clinics, the Seattle VA ICD clinics, Oregon Health and Sciences University ICD clinics and the Little Rock, Arkansas VA ICD clinics. Randomization and drug preparation were done by the Portland VA Medical Center research pharmacy. For safety purposes serum potassium will be measured at 1, 2, 3, 6, 12, 18, and 24 months. Patients will undergo ICD interrogation to document the occurrence of ICD therapy for VT or VF and will be screened for potential drug side effects every 3 months during the study. Health related quality of life will be measured at baseline, 3, 6, 12, 18, and 24 months using Short Form Health Survey adapted for veterans (SF36V) Veterans Health Study Version, the Patients Concerns Assessment, and the Kansas City Cardiomyopathy Questionnaire. Hospitalizations will be tracked throughout the study. In the subset of patient enrolled at the Portland VA the ventricular effective refractory period will be measured via single extra stimuli pacing through the ICD at 3 months after randomization.

ELIGIBILITY:
Inclusion Criteria:

-Patients were considered eligible for enrollment only if they had received

* an ICD therapy, either a shock or antitachycardia pacing (ATP),
* VT/VF in the previous 2 years or
* received an ICD for secondary prevention of sustained VT/VF in the previous 6 months.

Exclusion Criteria:

-Important exclusion criteria were

* an indication for spironolactone based on the RALES trial (EF of <35% and -New York Heart Association (NYHA) class III or IV),
* unstable angina,
* primary hepatic failure,
* known intolerance to spironolactone,
* a serum creatinine concentration of >2.5 mg/dL,
* a serum potassium concentration of >5.0 mmol/L, and
* a life expectancy of <2 years.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2004-07-28 (Actual); Primary Completion 2008-05-28 (Actual); Study Completion 2008-05-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Merritt Raitt, MD, Principal Investigator — VA Portland Health Care System, Portland, OR
Locations (1):
- VA Portland Health Care System, Portland, OR, Portland, Oregon, United States

IPD SHARING:
Plan to Share IPD: No
Patients did not give permission for data sharing

REFERENCES:
- [Result] Zarraga IG, Dougherty CM, MacMurdy KS, Raitt MH. The effect of spironolactone on ventricular tachyarrhythmias in patients with implantable cardioverter-defibrillators. Circ Arrhythm Electrophysiol. 2012 Aug 1;5(4):739-47. doi: 10.1161/CIRCEP.112.970566. Epub 2012 Jul 7. PMID 22773022
- [Derived] Liberato ACS, Raitt MH, Zarraga IGE, MacMurdy KS, Dougherty CM. Health-Related Quality of Life in the Spironolactone to Reduce ICD Therapy (SPIRIT) Trial. Clin Nurs Res. 2022 May;31(4):588-597. doi: 10.1177/10547738211036817. Epub 2021 Aug 6. PMID 34362264

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Spironolactone | Placebo
Started | 44 | 46
Completed | 44 | 46
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Spironolactone | Placebo | Total
Number analyzed (Participants) | 44 | 46 | 90
Age, Continuous [Mean (Standard Deviation); unit: years] | 66.6 (10.9) | 66.5 (9.3) | 66.5 (10.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 44 | 42 | 86
  Male | 0 | 4 | 4
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 44 | 46 | 90

OUTCOME MEASURES:

1. Primary Outcome: Time to First Appropriate Implantable Cardioverter Defibrillator (ICD) Therapy
Description: Time to first documented ICD therapy for ventricular tachycardia or ventricular fibrillation after randomization
Time Frame: through study completion, an average of 35 months
Population: all enrolled patients
Measure: Median (Full Range); unit: months
Arm/Group | Spironolactone | Placebo
Number analyzed (Participants) | 44 | 46
months | 8.8 [0 to 37.2] | 12.3 [0.3 to 38.5]
Statistical Analysis 1: Comparison: Spironolactone vs Placebo; Test type: Superiority; p = 0.71, Log Rank

2. Secondary Outcome: All Cause Hospitalization
Description: Number of patients hospitalized for any reason during study follow-up.
Time Frame: through study completion, an average of 35 months
Population: all randomized patients
Measure: Count of Participants; unit: Participants
Arm/Group | Spironolactone | Placebo
Number analyzed (Participants) | 44 | 46
Participants | 28 | 24
Statistical Analysis 1: Comparison: Spironolactone vs Placebo; Test type: Superiority; p = 0.07, Log Rank

3. Secondary Outcome: Ventricular Refractoriness
Description: The right ventricular effective refractory period (ERP) will be measured at 3 month in patients enrolled at the Portland VA Medical Center by single extra stimuli via their implanted defibrillator. The ERP is defined as the shortest paced beat coupling interval that fails to produce ventricular capture after a baseline stable pacing train.
Time Frame: measured 3 months after randomization
Population: Patients randomized at the Portland VA Hospital that consented to testing
Measure: Mean (Standard Deviation); unit: milliseconds
Arm/Group | Spironolactone | Placebo
Number analyzed (Participants) | 12 | 13
milliseconds | 294.2 (40.8) | 278.3 (24.1)
Statistical Analysis 1: Comparison: Spironolactone vs Placebo; Test type: Superiority; p = 0.42, t-test, 2 sided

4. Secondary Outcome: Short Form Health Survey Adapted for Veterans (SF36V)
Description: Short Form Health Survey adapted for veterans (SF36V) is a 36 item questionnaire that measures general physical and mental health [17]. The SF36V is a reliable and valid questionnaire, containing eight constructs of health status: physical functioning (PF), role limitations due to physical problems (RP), bodily pain (BP), general health perceptions (GH), energy/vitality (VT), social functioning (SF), role limitations due to emotional problems (RE), and mental health (MH). These eight dimensions can be summarized numerically into two scores, the physical component summary (PCS) and the mental component summary (MCS). Range 0-100 higher score is better Health Related Quality of Life (HRQOL). We are reporting the Mental Component Summary score at 12 months here.
Time Frame: 12 months after enrollment
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Spironolactone | Placebo
Number analyzed (Participants) | 44 | 46
score on a scale | 54.87 (22.50) | 63.31 (20.35)

5. Secondary Outcome: Patient Concerns Assessment (PCA)
Description: Patient Concerns Assessment (PCA) is a symptom checklist that measures physical symptoms and fears that are common after ICD implantation. The PCA is a disease-specific instrument for ICD QOL, symptoms, and distress, with a reliability of ( = 0.88). Range 0-44, a higher score reflects more concerns and fears.
Time Frame: 12 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Spironolactone | Placebo
Number analyzed (Participants) | 44 | 46
score on a scale | 22.15 (12.28) | 18.42 (10.06)

6. Secondary Outcome: Kansas City Cardiomyopathy Questionnaire (KCCQ)
Description: Kansas City Cardiomyopathy Questionnaire (KCCQ) is a 23-item reliable and valid questionnaire, which evaluates HRQOL in heart failure. It quantifies, in a disease-specific fashion, physical limitations, symptoms, quality of life, social interference and self-efficacy. KCCQ provides the calculation of 2 main scores, the overall score and the clinical summary score, which includes functional status, social limitation and quality of life domains scores. Range 0-100, higher scores represent higher HRQOL.
Time Frame: through study completion, an average of 35 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Spironolactone | Placebo
Number analyzed (Participants) | 44 | 46
score on a scale | 57.35 (28.59) | 68.67 (22.55)

ADVERSE EVENTS:
Time Frame: life of the study mean 35 months
Arm/Group | Spironolactone | Placebo
All-Cause Mortality (participants affected / at risk) | 13/44 | 12/46
Serious Adverse Events (participants affected / at risk) | 39/44 | 37/46
Other Adverse Events (participants affected / at risk) | 44/44 | 46/46
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Spironolactone (N=44) | Placebo (N=46)
hospitalization (General disorders) | 38 | 35 — hospitalization for any cause
death (General disorders) | 13 | 12
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Spironolactone (N=44) | Placebo (N=46)
Gynecomastia (Endocrine disorders) | 4 | 0
congestive heart failure (Cardiac disorders) | 34 | 33
Prerenal azotemia (Renal and urinary disorders) | 16 | 11
Any gastrointestinal issue (Gastrointestinal disorders) | 25 | 22

LIMITATIONS AND CAVEATS:
A limitation of this study was its small sample size. If a 35% relative risk reduction in the primary end point were assumed, the sample size of this trial would have given it 76% power with a type I error rate of 0.05.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No